CLINICAL TRIAL: NCT01509625
Title: Assessment of Treatment Response With Faslodex® (500 mg) in Standard Clinical Practice Through a Retrospective Study
Brief Title: Retrospective Study Assessment Treatment Response Faslodex®( 500 mg)
Acronym: EFFICACY
Status: Completed | Type: Observational
Sponsor: Isabel Blancas (Other)
Responsible Party: Sponsor-Investigator, Isabel Blancas, Medical Doctor, Hospital Clinico Universitario San Cecilio
Organization: Hospital Clinico Universitario San Cecilio (Other)
Other Study IDs: MIB-FUL-2011-01
Record Dates: First submitted 2011-12-29; First posted 2012-01-13 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2014-06

CONDITIONS: Malignant Neoplasm of Breast Stage IV
Keywords: Fulvestrant; Faslodex
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fulvestrant — It is an observacional retrospective study to asses the results of the administration of fulvestrant in the routine clinical practice.
  Other Names: Faslodex (registered)

SUMMARY:
This retrospective observational study is designed to assess the response to treatment with fulvestrant at a dose of 500 mg/month with a loading dose of 500 mg (LD-500), in terms of progression free survival (PFS), overall survival (OS), and clinical benefit rate (CBR), in post-menopausal women with Advanced Breast Cancer and estrogen receptor positive, who were treated with this medicinal product and at said dose after having progressed with a previous anti-estrogen therapy. During this study, a retrospective data collection will be carried out using the information contained in the Clinical History of said patients, provided that the treatment with fulvestrant at a dose of 500 mg and LD-500.

DETAILED DESCRIPTION:
Based on the results of the CONFIRM Study, a centralised change in the dosage of Faslodex® to 500 mg/month, with an additional pre-loading dose of 500 mg fourteen days after treatment smart was authorised in Europe; the dose is indicated for the treatment of post-menopausal women with ABC, hormone receptor positive and whose disease had progressed after anti-estrogen therapy.

Several sites worldwide participated in this study, but given the importance of the results obtained and their impact, we believe it is important to have local data available in Spain that would enable us to determine how this new 500 mg dose of Faslodex® behaves in the treatment and to assess treatment response within standard clinical practice and the current indications of this drug.

Therefore, we designed this retrospective, observational study in which we will measure response in term of PFS using data collected from the Clinical History.

Likewise, other variables will be studied: OS, CBR, duration of clinical benefit, tolerability and safety. Patient subgroups, like those who over-express her-2, according to levels of ki-67 and the presence or not of visceral metastases will also be studied.

This retrospective observational study is designed to assess the response to treatment with fulvestrant at a dose of 500 mg/month with a loading dose of 500 mg (LD-500), in terms of progression free survival (PFS), overall survival (OS), clinical benefit rate (CBR), and duration of clinical benefit (DCB, in post-menopausal women with Advanced Breast Cancer and estrogen receptor positive, who were treated with this medicinal product and at said dose after having progressed with a previous anti-estrogen therapy. During this study, a retrospective data collection will be carried out using the information contained in the Clinical History of said patients, provided that the treatment with fulvestrant at a dose of 500 mg and LD-500, had occurred at some point between 1 January 2010 and 31 October 2011 (hereinafter, the study period).

Thus, we will obtain the PFS, OS and CBR data, as well as information on safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent from patients when possible.
* In the event of patients who are deceased at the time of inclusion, no signed informed consent will be available; thus, the investigator assumes the responsibility of data protection and confidentiality and of safeguarding the processing of the data.
* Post-menopausal women.
* Diagnosed with locally advanced or Metastatic Breast Cancer with histological/cytological confirmation.
* Documented estrogen receptor positive status for the primary tumour.
* Patient who, after progression with a previous anti-estrogen treatment, received treatment at some time with fulvestrant (Faslodex®) at the 500 mg/month and LD-500 dose during the study period.

Exclusion Criteria:

* Having received treatment with unapproved or experimental drugs during the study period.
* Presenting another concomitant cancer other than stage I cervical cancer or cutaneous tumours without lymph node or distant involvement.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-menopausal women with Advanced Breast Cancer (ABC) and estrogen receptor positive (ER+) who were treated with this medicinal product and at said dose after having progressed with a previous anti-estrogen therapy
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Blancas, MD, Principal Investigator
Locations (7):
- Spain (7):
  - Hospital San Cecilio, Granada, Granada
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital Torrecardenas Almería, Almería
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital SAS Jeréz de la Frontera, Jeréz de La Frontera
  - Hospital Costa del Sol, Marbella
  - Hospital Carlos Hayas, Málaga

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- One Arm of Metastatic Breast Cancer Patients: All the patients have tumors with positive estrogen receptors
Period: Overall Study
Arm/Group | One Arm of Metastatic Breast Cancer Patients
Started | 272
Completed | 263
Not Completed | 9

BASELINE CHARACTERISTICS:
Groups:
- One Arm of Metastatic RE Breast Cancer Patients: Women with metastatic breast cancer who have disease progresion after prior antiestrogen treatment. All tumors were positive estrogen receptors
Arm/Group | One Arm of Metastatic RE Breast Cancer Patients
Number analyzed (Participants) | 272
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 134
  >=65 years | 138
Age, Continuous [Mean (Full Range); unit: years]
  age | 65 [64.2 to 67.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272
  Male | 0
Region of Enrollment [Number; unit: participants]
  Spain | 272
Histologic type [Number; unit: participants]
  ductal | 208
  lobulillar | 37
  ductal+lobulillar | 7
  others | 7
  not known | 13
Estrogen receptor and Progesterone receptor status [Number; unit: participants]
  ER positive and PGR positive | 197
  ER positive and PGR negative | 61
  ER negative and PGR positive | 1
  No specifical information | 13

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Response to treatment with fulvestrant (Faslodex®) in terms of Progression Free Survival.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% or more increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 22 months
Measure: Median (95% Confidence Interval); unit: month
Groups:
- One Arm of Metastatic Breast Cancer Patients: All patients have tumors with positive estrogen receptors
Arm/Group | One Arm of Metastatic Breast Cancer Patients
Number analyzed (Participants) | 263
month | 10.6 [9.0 to 11.5]

2. Secondary Outcome: Clinical Benefit Rate
Description: Response to treatment with fulvestrant in terms of Clinical Benefit Rate. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or TC: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; PD (progressive disease)> = 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion or the appearance of new lesions; Clinical Benefit = CR + PR+ Stable Disease (not progression of the disease for 24 or more weeks).
Time Frame: 22 months
Measure: Number; unit: percentage of patients
Arm/Group | One Arm of Metastatic Breast Cancer Patients
Number analyzed (Participants) | 263
percentage of patients | 56.5

3. Secondary Outcome: Overall Survival
Description: Response to treatment with fulvestrant in terms of Overall Survival
Time Frame: 22 months
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | One Arm of Metastatic Breast Cancer Patients
Number analyzed (Participants) | 263
month | 43.2 [37.0 to 49.2]

4. Secondary Outcome: Duration of Clinical Benefit
Description: Response to treatment with fulvestrant in terms of Duration of the Clinical Benefit.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or TC: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; PD (progressive disease)> = 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion or the appearance of new lesions; Clinical Benefit = CR + PR+ Stable Disease (not progression of the disease for 24 or more weeks).
Time Frame: 22 months
Population: For the study of the duration of the clinical benefit, only the patients that get a clinical benefit could be analyzed (this is the reason becasuse the number of participants analyzed was 140)
Measure: Median (95% Confidence Interval); unit: month
Groups:
- Patients With Clinical Benefit: Patients wich achieved a clinical benefit with fulvetrant 500: complete response, partial response or stable disease of 24 weeks or longer
Arm/Group | Patients With Clinical Benefit
Number analyzed (Participants) | 140
month | 18.4 [14.5 to 23.0]

5. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: 22 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | One Arm of Metastatic Breast Cancer Patients
Number analyzed (Participants) | 263
percentage of patients
  any toxicity | 35.4 [29.6 to 41.5]
  local pain injection | 9.9 [6.6 to 14.1]
  Muscle-bone pain | 7.2 [4.4 to 11.1]
  Gastrointestinals disorders | 6.8 [4.1 to 10.6]
  Hot flashes | 6.1 [3.5 to 9.7]
  Urinary infection | 0.8 [0.1 to 2.7]
  Weight gain | 0.8 [0 to 2.1]
  Vaginitis | 0.4 [0 to 2.1]
  Joint pain | 16 [11.8 to 21]

6. Secondary Outcome: Response to Treatment With Fulvestrant in Terms of PFS in a Subgroup of Patients With Visceral Metastases and Without Visceral Metastases
Description: Response to treatment with fulvestrant at the 500 mg/month and LD 500 dose in terms of PFS in a subgroup of patients with visceral metastases and without visceral metastases.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or TC: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; PD (progressive disease)> = 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion or the appearance of new lesions; Clinical Benefit = CR + PR+ Stable Disease (not progression of the disease for 24 or more weeks).
Time Frame: 22 months
Population: We identified 272 patientes for the study but nine subjects were ineligible due to lack of information, leaving to 263 evaluable patients.
Measure: Median (95% Confidence Interval); unit: month
Groups:
- Patients Without Visceral Metastasis: Group of patients without metastasis in organs like liver or lungs
- Patients With Visceral Metastasis: Group of patients with metastasis in organs like liver or lungs
Arm/Group | Patients Without Visceral Metastasis | Patients With Visceral Metastasis
Number analyzed (Participants) | 225 | 38
month | 10.6 [8.9 to 10.6] | 10 [7.1 to 13.9]

7. Secondary Outcome: Response to Treatment With Fulvestrant in Terms of PFS in a Subgroup of Patients After a First-line Hormonal Therapy Prior and in Subgroup of Patients After Two or More Prior Lines of Hormonal Therapy
Description: To assess the response to treatment with fulvestrant (Faslodex®) at the 500 mg/month and LD-500 dose in terms of PFS in a subgroup of patients after a first-line hormonal therapy prior and in subgroup of patients after two or more prior lines of hormonal therapy
Time Frame: 22 months
Population: We identified 272 patientes for the study but nine subjects were ineligible due to lack of information, leaving to 263 evaluable patients. There were 5 patients that have not received previous tamoxifen or an aromatases inhibitor, so they are not included in one of these two groups.
Measure: Median (95% Confidence Interval); unit: month
Groups:
- Previous Treatment Wiht One Line of Hormonal Treatment: Hormonal treatment was tamoxifen or an aromatase inhibitor
- Previous Treatment With Two or More Hormonal Treatment Lines: The patients have received at least two hormonal treatment: tamoxifen and aromatase inhibitor
Arm/Group | Previous Treatment Wiht One Line of Hormonal Treatment | Previous Treatment With Two or More Hormonal Treatment Lines
Number analyzed (Participants) | 128 | 130
month | 11.2 [9.5 to 13.6] | 9.2 [7.4 to 11.2]

8. Secondary Outcome: Response to Treatment With Fulvestrant in Terms of PFS in Subgroups of Patients With Her-2 Overexpression and Those Who do Not Over-express Her-2
Description: To assess the response to treatment with fulvestrant at the 500 mg/month and LD 500 dose in terms of PFS in subgroups of patients with her-2 overexpression (+++ by immunohistochemistry or FISH positive) and those who do not over-express her-2 and to compare both groups.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or TC: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; PD (progressive disease)> = 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion or the appearance of new lesions; Clinical Benefit = CR + PR+ Stable Disease (not progression of the disease for 24 or more weeks).
Time Frame: 22 months
Population: We identified 272 patientes for the study but nine subjects were ineligible due to lack of information, leaving to 263 evaluable patients. There were no information regarding HER2 status in 31 patients.
Measure: Median (95% Confidence Interval); unit: month
Groups:
- Patients With Tumors HER2 Positive: tumor is considered HER2 positive if there is a sobreexpression of the receptor by immunohistochemistry or FISH is positive
- Patients With Tumors HER2 Negative: tumor is considered HER2 negative if there is not a sobreexpression of the receptor by immunohistochemistry or FISH is positive
Arm/Group | Patients With Tumors HER2 Positive | Patients With Tumors HER2 Negative
Number analyzed (Participants) | 26 | 206
month | 10.2 [7.7 to 13.3] | 10.3 [8.0 to 11.3]

9. Secondary Outcome: Response to Treatment With Fulvestrant in Terms of PFS in a Subgroup of Patients With Elevated Ki-67 and With Low Ki-67
Description: To assess the response to treatment with fulvestrant (Faslodex®) at the 500 mg/month and LD-500 dose in terms of PFS in a subgroup of patients with elevated ki-67 (greater than or equal to 20%) and with low ki-67 and to compare both groups
Time Frame: 22 months
Population: We identified 272 patientes for the study but nine subjects were ineligible due to lack of information, leaving to 263 evaluable patients. There were no information regarding tumor ki67 expresion in 121 patients.
Measure: Median (95% Confidence Interval); unit: month
Groups:
- Patients With Tumors ki67 Positive: Patients with tumors with high ki67 expression
- Patients With Tumors ki67 Negative: Patients with tumors with low ki67 expression
Arm/Group | Patients With Tumors ki67 Positive | Patients With Tumors ki67 Negative
Number analyzed (Participants) | 70 | 72
month | 9.6 [6.5 to 13.1] | 10.0 [7.8 to 12.9]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | One Arm of Metastatic Breast Cancer Patients
Serious Adverse Events (participants affected / at risk) | 0/263
Other Adverse Events (participants affected / at risk) | 93/263
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | One Arm of Metastatic Breast Cancer Patients (N=263)
Gastrointestinal disorders (Gastrointestinal disorders) | 18
Pain in inyection site (Injury, poisoning and procedural complications) | 26
Musculoskeletal disorders (Musculoskeletal and connective tissue disorders) | 19
Hot flushes (Skin and subcutaneous tissue disorders) | 16
Urinary infection (Infections and infestations) | 2
Weight gain (Endocrine disorders) | 1
Vaginitis (Infections and infestations) | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No